CLINICAL TRIAL: NCT04019353
Title: Cf-DNA Assay During Treatment of Acute Rejection-Pilot Study
Brief Title: Cf-DNA Assay During Treatment of Acute Rejection
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: SURG-2018-27247
Record Dates: First submitted 2019-06-21; First posted 2019-07-15 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Kidney Transplant Failure and Rejection; Kidney Transplant; Complications; Kidney Transplant Rejection; Transplant; Complication, Rejection; Transplant Dysfunction
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cf-DNA Collection: All patients undergoing kidney allograft biopsy for suspicion of an acute rejection episode will be approached for consent into the study. Patients who consent to the study will have the cf-DNA test drawn at time of biopsy to determine levels of cf-DNA. All consented patients will be followed for biopsy outcomes. Those whose biopsy shows acute rejection leading to treatment will have cf-DNA determination at 2, 4, 6, and 8 weeks post biopsy. Recipients with persistent high cf-DNA levels will undergo repeat biopsy at ~6 weeks after end of treatment per standard of care (this is not performed for purpose of the study, but for clinical care).
  Interventions: Genetic: cf-DNA Collection

INTERVENTIONS:
Genetic: cf-DNA Collection — For all consenting recipients undergoing kidney biopsy between 1 and 12 months post-transplant, a single tube of blood will be drawn (at the time of other blood draws so that there is no additional needle stick) to measure cf-DNA. The tube will be shipped to the California lab for determination of donor cf-DNA. For recipients whose biopsy shows AR, a tube of blood will be drawn at 2, 4, 6, and 8 weeks after initiation of anti-rejection treatment and similarly will be shipped to the California lab for determination of cf-DNA.
  Recipients whose exit biopsy shows ongoing inflammation and receiving additional anti-rejection therapy will have an additional exit biopsy additional cf-DNA determinations.

SUMMARY:
The objective of this study is to determine whether cell-free DNA (cf-DNA) measurement can be used as a biomarker for successful treatment of an acute rejection (AR) episode after kidney transplantation.

A fall in donor cf-DNA level may be a biomarker for successful AR treatment. The goal is to do an exploratory study to determine, in recipients with biopsy-proven AR, whether persistence or elevated levels of donor cf-DNA are associated with ongoing inflammation at the time of exit biopsy; and whether fall in donor cf-DNA level is associated with successful AR treatment.

Measurement of cf-DNA has recently been started for kidney transplant recipients. There will be two groups of patients eligible for this study:

1. those who have had sequential measurement of cf-DNA prior to graft dysfunction leading to a biopsy, and
2. those who have not had previous measurement of cf-DNA

DETAILED DESCRIPTION:
Significance of Research Question/Purpose:

A kidney transplant biopsy is the gold standard for making a diagnosis at the time of graft dysfunction. However, there are risks associated with a transplant biopsy (e.g., hematuria, clots within the collecting system, bleeding, hematoma within the kidney, urine leak, and rarely AKI and/or graft loss). Recently, a blood test has been developed which distinguishes donor and recipient circulating cf-DNA. Using this methodology, circulating cf-DNA is amplified, then using a panel of markers, 2 DNA peaks can be observed - a high peak for the recipient DNA and a very low peak for the donor (importantly, this is not genetic testing; only high and low peaks are identified). When cf-DNA is measured at the time of a kidney biopsy for graft dysfunction, an elevated donor cf-DNA level - compared to that seen in a cohort without inflammation - can be seen in recipients with an acute rejection (AR) episode. Data, to date, suggests that if >1% of cf-DNA is donor derived, there is likely graft inflammation.

Currently, there are ongoing studies to determine if sequential measurement of cf-DNA in the same recipient will show elevated donor cf-DNA levels earlier than a serum creatinine rise, thus potentially allowing earlier detection and treatment of AR episodes.

Serum creatinine level is used as a marker for successful treatment of an acute rejection episode. However, creatinine level is an insensitive marker of response to treatment of both cellular and antibody mediated rejection. Studies in which biopsies are done at the end of "presumed" successful rejection treatment show that some patients whose creatinine level returned to baseline have ongoing inflammation. Unless additional anti-rejection treatment is given, this incomplete treatment leads to increased risk for donor-specific antibody formation and graft failure.

As a consequence, the investigators (the U of MN Kidney Transplant Program) are now doing routine "exit" biopsies for patients treated for acute rejection episodes and whose serum creatinine level returns to baseline. The investigators have always done biopsies in patients whose creatinine level did not return to baseline. The "exit" biopsy is done at ~6 weeks after completion of rejection treatment. If the exit biopsy shows ongoing inflammation, additional rejection treatment is considered.

It would be ideal to have a noninvasive marker for successful rejection treatment. The objective of this study is to determine whether cell-free DNA (cf-DNA) measurement can be used as a biomarker for successful treatment of an acute rejection (AR) episode after kidney transplantation.

The addition of cf-DNA testing would have two potential benefits:

1. Serum creatinine may return to baseline (pre-rejection level), but ongoing allograft injury may be occurring as creatinine is an insensitive marker of subtle allograft dysfunction. This inflammation is known to create antigenic presentation that results in DSA production which is major cause of long-term allograft loss
2. Serum creatinine may not return to baseline as there is irreparable allograft loss or intensification of CNI dosing. This would result in a biopsy that does not change management, but would put the patient through an unnecessary and potentially harmful procedure. If a non-invasive marker decreases with treatment and correlates with complete resolution of rejection episode, this would be useful for monitoring purposes.

Preliminary Data:

1. The University of MN Transplant Program participated in the original studies showing an association between cf-DNA and acute rejection. The investigators have experience with the methodology and with working with the company that does the cf-DNA assay
2. Since starting to do exit biopsies the investigators, like others, have found that some patients with presumed successful rejection treatment have evidence of ongoing inflammation seen in the biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant recipients undergoing transplant biopsy between 1 and 12 months post-transplant because of graft dysfunction.

Exclusion Criteria:

* <1 months post-transplant
* >12 months post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients undergoing transplant biopsy between 1 and 12 months post-transplant because of graft dysfunction.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Number of participants converted to <1% measured donor cf-DNA concentrations | 8 weeks
  Number of patients with donor cf-DNA >1% who achieve an intra-patient change of measured donor cf-DNA to less than 1% from the time of kidney biopsy for AR to 6 weeks after initiation of treatment.
Number of participants who achieve 61% reduction in measured donor cf-DNA concentrations | 8 weeks
  Number of patients who do not have > 1% donor cf-DNA at the time of rejection who achieve a reduction in donor cf-DNA by 61%.

SECONDARY OUTCOMES:
Number of participants who return to baseline measured donor cf-DNA concentrations | 8 weeks
  Number of patients for whom a baseline of donor cf-DNA has been ascertained through monitoring prior to acute rejection and who return to baseline cf-DNA after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No